CLINICAL TRIAL: NCT00546195
Title: Expression Profiling of Bacterial Lipopolysaccharide Activated Neutrophil in Pre-Term, Term Infants and Adults
Brief Title: Infant Immune Response to Bacterial Infection
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999908011; 08-CH-N011
Record Dates: First submitted 2007-10-17; First posted 2007-10-18 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-03-29

CONDITIONS: Prematurity; Histologic Chorioamnionitis
Keywords: Cord Blood; Neutrophils; Polysaccharide; Gene Expression
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will examine the response of white blood cells to bacterial infection in blood taken from the umbilical cords of newly delivered infants. The blood samples will be taken from both male infants who were carried to term and male infants who were born prematurely, and genetic studies will compare these blood samples to samples drawn from healthy adult male volunteers. The study is designed to look at the ways in which the immune systems of newborn infants respond to bacterial infection.

Participants in this study will be pregnant Chinese women admitted to the labor ward of the Prince of Wales Hospital (Sha Tin district of New Territories, Hong Kong SAR) for normal spontaneous delivery. Those with known blood-borne infectious diseases such as HIV and hepatitis B will be excluded from this study.

Cord blood and placenta samples will be collected after the completion of delivery. The samples collected for this study will be restricted to male newborns. A comparison group of blood samples will be drawn from healthy male adults between 25 and 35 years of age....

DETAILED DESCRIPTION:
Bacterial infection in preterm neonates is a significant clinical problem. Neutrophils play a critical role in the bactericidal process, which is immature in newborns though their peripheral blood neutrophil counts are similar to or higher than that of older children and adults. The use of steroids to enhance lung maturation in premature infants complicates this problem. Many studies have shown different biological activities between lipopolysaccharide (LPS) activated neonatal cord blood neutrophils and adult peripheral blood neutrophils. In spite of a number of previous studies, the genetic basis of this differential response to LPS-activation remains unknown. In this study, we will identify the differential gene expression profiles of LPS-activated adult peripheral blood versus cord blood neutrophils from both term and preterm infants by whole genome ligonucleotide microarray. We will investigate the priming effect of histologic chorioamnionitis (HCA), a severe infection/inflammation implicated in many neonatal diseases, on the immune response in neutrophils in terms of gene expression. The effect of prenatal administration of steroids on the immune response in preterm neutrophils is another question we will address in the proposed study. This study will provide insight into the molecular basis for genetic regulation of neutrophil development. We expect to identify novel genes with differential expressions in LPS-activated cord blood neutrophils when compared to those of LPS-activated adult cells. Aberrant transcripts due to the priming effect of HCA to the immune response in term neutrophils will also provide insight on the defense mechanism of subsequent exposures to bacterial infection.

This is a collaborative study. All samples will be collected by our Collaborators at the Chinese University of Hong Kong, Hong Kong. We will perform expression profiling in the Laboratory of Clinical Genomics at NICHD. This protocol has been approved by the Joint Clinical Research Ethics Committee of the Chinese University of Hong Kong and Hospital Authority of Hong Kong.

ELIGIBILITY:
* INCLUSION CRITERIA:

Chinese pregnant women admitted to the labor ward of the Prince of Wales hospital.

Normal spontaneous delivery.

EXCLUSION CRITERIA:

Patient diagnosed with known infectious diseases such as HIV and HBV positive cases (blood precautions).

Patients are incompetent to consent such as being mentally retarded or mentally ill and without an impairment of judgment at the time of consenting.

Patients who do not consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2007-10-15; Study Completion 2011-03-29

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Child Health and Human Development (NICHD), 9000 Rockville, Bethesda, Maryland, United States

REFERENCES:
- [Background] Fanaroff AA, Korones SB, Wright LL, Verter J, Poland RL, Bauer CR, Tyson JE, Philips JB 3rd, Edwards W, Lucey JF, Catz CS, Shankaran S, Oh W. Incidence, presenting features, risk factors and significance of late onset septicemia in very low birth weight infants. The National Institute of Child Health and Human Development Neonatal Research Network. Pediatr Infect Dis J. 1998 Jul;17(7):593-8. doi: 10.1097/00006454-199807000-00004. PMID 9686724
- [Background] Kylat RI, Ohlsson A. Recombinant human activated protein C for severe sepsis in neonates. Cochrane Database Syst Rev. 2006 Apr 19;(2):CD005385. doi: 10.1002/14651858.CD005385.pub2. PMID 16625638
- [Background] Gladstone IM, Ehrenkranz RA, Edberg SC, Baltimore RS. A ten-year review of neonatal sepsis and comparison with the previous fifty-year experience. Pediatr Infect Dis J. 1990 Nov;9(11):819-25. doi: 10.1097/00006454-199011000-00009. PMID 2263432